CLINICAL TRIAL: NCT04284618
Title: Off Axis View Radiographs Assessing Hallux Valgus Interphalangeus in Hallux Valgus Deformity: A Comparison With the Traditional Anteroposterior Standing Radiographs
Brief Title: Off Axis View Radiographs Assessing Hallux Valgus Interphalangeus in Hallux Valgus Deformity
Status: Completed | Type: Observational
Sponsor: Dr.Gerhard Kaufmann (Other)
Collaborators: Medical University Innsbruck (Other)
Responsible Party: Sponsor-Investigator, Dr.Gerhard Kaufmann, Dr. Gerhard Kaufmann, Principal investigator and Head of the Orthopaedic and Foot Center Innsbruck, OFZ Innsbruck
Organization: OFZ Innsbruck (Other)
Other Study IDs: 1100/2019
Record Dates: First submitted 2020-02-19; First posted 2020-02-26 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Hallux Valgus Interphalangeus; Hallux Valgus
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- assessment of radiographic angles on standardized films: On Standing standardized radiographs of the foot the most common angles for describing a hallux valgus interphalangeus deformity are measured. The measured angles are the following: The hallux interphalangeal angle (HIA), the proximal to distal phalangeal articular angle (PDPAA), the proximal phalangeal articular angle (PPAA) or distal articular set angle (DASA), and the distal phalangeal articular angle (DPAA).
  Interventions: Diagnostic Test: assessment of standardized and off axis view radiographs
- assessment of radiographic angles on off axis view films: On off axis view radiographs of the foot the most common angles for describing a hallux valgus interphalangeus deformity are measured. The measured angles are the following: The hallux interphalangeal angle (HIA), the proximal to distal phalangeal articular angle (PDPAA), the proximal phalangeal articular angle (PPAA) or distal articular set angle (DASA), and the distal phalangeal articular angle (DPAA).
  Interventions: Diagnostic Test: assessment of standardized and off axis view radiographs

INTERVENTIONS:
Diagnostic Test: assessment of standardized and off axis view radiographs — Radiographic assessment of hallux valgus interphalangeus angles is performed on preoperative standing anteroposterior and on off axis view radiographs. These radiographs are taken by equalizing the hyperpronation of the greater toe.

SUMMARY:
In hallux valgus deformity an additional deformity of the proximal phalangeal bone can be observed frequently as well. Due to a hyperpronation of the greater toe on standardized radiographs the deformity defining angles are likely to be underestimated. Therefore the investigators developed an off axis view radiograph for determining the real deformity. This study compares the standardized and the off axis view radiographs.

DETAILED DESCRIPTION:
Hallux valgus is a frequent deformity of the first ray of the foot with adduction and pronation of the greater toe at the first metatarsophalangeal joint and abduction of the first metatarsal at the first tarsometatarsal joint. Valgus deformity of the greater toe itself - so called "Hallux valgus interphalangeus (HVI)" - can be found regularly in hallux valgus deformities as well. Various osteotomies and soft tissue procedures to correct hallux valgus deformity have been proposed so far. While corrective osteotomies of the first metatarsal bone represent the main therapeutical option in hallux valgus correction, the need for additional phalangeal osteotomy of the greater toe (e.g., Akin osteotomy) is discussed controversial and remains a surgeon's decision to date. In this context, the decision to perform an additional Akin osteotomy depends on the radiographic measurement of the hallux valgus interphalangeus deformity.

The following radiographic angles to define HVI have been used most consistently in the literature so far: The hallux interphalangeal angle (HIA), the proximal to distal phalangeal articular angle (PDPAA), the proximal phalangeal articular angle (PPAA) or distal articular set angle (DASA), and the distal phalangeal articular angle (DPAA). To date, a hallux valgus interphalangeal angle of greater than 10 degrees serves as the most frequently used definition of HVI. However, the measurement of HIA is prone to error due to the irregular geometry of the distal phalanx. Therefore, the proximal to distal phalangeal articular angle might describe hallux valgus interphalangeus deformity more precisely and reliably. Furthermore, a significant hyperpronation of the phalangeal bone can be observed frequently in hallux valgus deformity. This phalangeal hyperpronation results in a non-orthogonal projection of the greater toe on preoperative films, which might be the cause for underestimation of HVI on standardized weightbearing radiographs.

The aim of this study is to investigate the reliability of radiological assessment of hallux valgus interphalangeus and to evaluate, if HVI can be defined more precisely using intraoperative anteroposterior "off axis view" radiographs additionally. The investigators hypothesize that (1) HVI is underestimated on pre-operative standardized anteroposterior radiographs compared to anteroposterior off axis views; (2) the Investigators hypothesize that PDPAA shows significantly less intra- and interobserver variance and is therefore more reliable than other angles (HIA, PPAA, DPAA) for measuring HVI; and (3) the investigators hypothesize, that the detected differences between weightbearing and off axis radiographs are a function of the severity of the deformity

ELIGIBILITY:
Inclusion Criteria:

* All patients who have undergone surgery for hallux valgus deformity by open or minimally invasive percutaneous hallux valgus correction at the Orthopedic and Foot Center Innsbruck between November 2018 and May 2019.

Exclusion Criteria:

* Incomplete radiological data (preoperative and intraoperative radio-graphs)
* Pregnancy
* missing of written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: a retrospective cohort of 60 patients is assessed
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-11-10 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
reliability of standardized Standing radiographs for defining hallux valugs interphalangeus | 12 weeks
  Analysis of the reliability of radiological angles hallux valgus interphalangeus and evaluation, if Hallux valgus interphalangeus can be determined more precisely on off axis view radiographs. Evaluation is made with specific radiographic angles. The used angles are the following: hallux interphalangeal angle (HIA), the proximal to distal phalangeal articular angle (PDPAA), the proximal phalangeal articular angle (PPAA) or distal articular set angle (DASA), and the distal phalangeal articular angle (DPAA).

SECONDARY OUTCOMES:
correlation of hallux valgus interphalangeus angles with the severity of hallux valgus deformity | 12 weeks
  analysis of hallux valgus severity and ist influence on weightbearing and off axis radiographs by the use of radiographic angles. The used angles are the following: hallux interphalangeal angle (HIA), the proximal to distal phalangeal articular angle (PDPAA), the proximal phalangeal articular angle (PPAA) or distal articular set angle (DASA), and the distal phalangeal articular angle (DPAA).

CONTACTS AND LOCATIONS:
Locations (1):
- Gerhard Kaufmann, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaufmann G, Sinz S, Giesinger JM, Braito M, Biedermann R, Dammerer D. Loss of Correction After Chevron Osteotomy for Hallux Valgus as a Function of Preoperative Deformity. Foot Ankle Int. 2019 Mar;40(3):287-296. doi: 10.1177/1071100718807699. Epub 2018 Oct 31. PMID 30379084
- [Background] Partio N, Maenpaa H, Huttunen T, Haapasalo H, Laine HJ, Mattila VM. Incidence of hallux valgus primary surgical treatment. Finnish nationwide data from 1997 to 2014. Foot Ankle Surg. 2019 Dec;25(6):761-765. doi: 10.1016/j.fas.2018.10.001. Epub 2018 Oct 17. PMID 31796164
- [Background] Deenik A, van Mameren H, de Visser E, de Waal Malefijt M, Draijer F, de Bie R. Equivalent correction in scarf and chevron osteotomy in moderate and severe hallux valgus: a randomized controlled trial. Foot Ankle Int. 2008 Dec;29(12):1209-15. doi: 10.3113/FAI.2008.1209. PMID 19138485
- [Background] Klugarova J, Hood V, Bath-Hextall F, Klugar M, Mareckova J, Kelnarova Z. Effectiveness of surgery for adults with hallux valgus deformity: a systematic review. JBI Database System Rev Implement Rep. 2017 Jun;15(6):1671-1710. doi: 10.11124/JBISRIR-2017-003422. PMID 28628523
- [Background] Thordarson DB, Rudicel SA, Ebramzadeh E, Gill LH. Outcome study of hallux valgus surgery--an AOFAS multi-center study. Foot Ankle Int. 2001 Dec;22(12):956-9. doi: 10.1177/107110070102201205. PMID 11783920
- [Background] Kaufmann G, Hofmann M, Braito M, Ulmer H, Brunner A, Dammerer D. Need for concomitant Akin osteotomy in patients undergoing Chevron osteotomy can be determined preoperatively: a retrospective comparative study of 859 cases. J Orthop Surg Res. 2019 Aug 28;14(1):277. doi: 10.1186/s13018-019-1319-2. PMID 31455364
- [Background] Kaufmann G, Hofmann M, Ulmer H, Putzer D, Hofer P, Dammerer D. Outcomes after scarf osteotomy with and without Akin osteotomy a retrospective comparative study. J Orthop Surg Res. 2019 Jun 26;14(1):193. doi: 10.1186/s13018-019-1241-7. PMID 31242910